CLINICAL TRIAL: NCT00047931
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Multiclade HIV-1 DNA Plasmid Vaccine, VRC-HIVDNA009-00-VP in Uninfected Adult Volunteers
Brief Title: HIV-1 Vaccine Test in Uninfected Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030022; 03-I-0022
Record Dates: First submitted 2002-10-22; First posted 2002-10-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-05-05

CONDITIONS: HIV Seronegativity; AIDS Vaccines
Keywords: Healthy; HIV-Negative; Placebo-Controlled; Volunteer; Dose-Escalation; HIV Seronegativity; Healthy Volunteer; HV

INTERVENTIONS:
Drug: VRC-HIVDNA009-00-VP

SUMMARY:
This study will test the safety of an experimental vaccine against HIV and examine whether it induces an immune response to HIV. A vaccine is a substance given to try to create resistance or immunity to a disease or infection. The vaccine in this study is made from DNA (genetic material) of four HIV proteins called 'gag', 'pol', 'Nef', and 'Env'. Injected into a human, the viral DNA instructs the body to make small amounts of some HIV proteins. This study will see if the body then creates an immune response to these proteins. Study participants cannot catch HIV or AIDS from the DNA vaccine or any proteins made from it.

Healthy normal volunteers between 18 and 40 years of age may be eligible for this study. Candidates will be screened with a medical history, physical examination and blood and urine tests. Women will also have a pregnancy test. Women enrolled in the study must either be infertile (e.g., due to menopause or hysterectomy) or must agree either to abstain from heterosexual sex or to practice birth control for at least 21 days before beginning the study and throughout its duration.

Participants will be randomly assigned to receive either the experimental vaccine or a placebo (a salt solution that does not contain any active substance) and will be divided into three groups, based on their entry into the study. Of the first seven people enrolled (Group 1), five will receive a 2-mg dose of vaccine and two will receive placebo. If the vaccine is safe at this dose, then in Group 2, five people will receive a 4-mg dose of vaccine and two will receive placebo. If this dose is safe, then in Group 3, thirty people will receive an 8-mg dose of vaccine and six will receive placebo.

All participants will receive three injections in an upper arm muscle-one injection a month for three months-with a needle-less device called a Biojector 2000® (Registered Trademark). At the time of each injection, participants will be observed for at least 1 hour after immunization. At home, they will record their temperature and any symptoms they may experience, including any effects at the injection site, for at least 7 days, or as long as the symptoms remain. If symptoms occur, participants will report them immediately to the clinic staff and, if necessary, come to the clinic for an examination.

Participants will have about 10 clinic visits during the study. Most visits will last about 2 hours; those on vaccination days will last about 4 hours. ...

DETAILED DESCRIPTION:
This is a Phase I, randomized, controlled, double-blinded, dose-escalation study to examine tolerability, dose, and immune response of an HIV DNA plasmid vaccine. The hypothesis is that this vaccine will be safe for human administration and elicit immune responses to HIV. The primary objective is to evaluate the safety and tolerability in humans of VRC-HIVDNA009-00-VP and secondary objectives are to evaluate the immunogenicity of the vaccine and social impact of participating in an HIV-1 vaccine trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

* 18 to 40 years old.
* Available for follow-up for the duration of the study (12 months).
* Able to provide proof of identity to the acceptance of the study clinician completing the enrollment process.
* Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.
* Able and willing to sign the informed consent form.
* Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.
* Willing to have blood samples used for future research.
* Willing to discuss HIV infection risks and amenable to risk reduction counseling.
* In good general health without clinically significant medical history.
* Physical examination and laboratory results without clinically significant findings within the 28 days prior to enrollment.

Laboratory Criteria within 28 days prior to enrollment:

* Hematocrit greater than or equal to 34 percent for women; greater than or equal to 38 percent for men.
* WBC count: Non-African Americans equals 3,300-12,000 cells/mm(3); African-Americans equals 2,500-12,000 cells/mm(3) (in the absence of clinical or pathological etiology).
* Differential either within institutional normal range or accompanied by site physician approval.
* Total lymphocyte count: Non-African Americans greater than or equal to 800 cells/mm(3); African Americans greater than or equal to 650 cells/mm(3) (in the absence of clinical or pathological etiology).
* Platelets equals 125,000-550,000/mm(3).
* ALT (SGPT) less than or equal to 1.5 times upper limit of normal.
* Serum creatinine less than or equal to 1.3 mg/dL.
* Normal urinalysis defined as negative glucose, negative or trace protein, and negative or trace hemoglobin (blood).
* Negative FDA-approved HIV blood test.
* Negative Hepatitis B surface antigen.
* Negative anti-HCV or negative HCV PCR if the anti-HCV is positive.

Female-Specific Criteria:

* Negative beta-HCG pregnancy test for women presumed to be of reproductive potential.
* A female participant must meet one of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

Or

-Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and throughout the duration of the study,

Or

* Participant agrees to consistently practice contraception at least 21 days prior to enrollment and throughout the duration of the study by one of the following methods:
* condoms, male or female, with or without a spermicide.
* diaphragm or cervical cap with spermicide.
* intrauterine device.
* contraceptive pills, Norplant, or Depo-Provera.
* male partner has previously undergone a vasectomy for which there is documentation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

-Woman who is breast-feeding.

Volunteer has received any of the following substances:

* HIV vaccines in a prior clinical trial.
* Immunosuppressive or cytotoxic medications within the past six months with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis.
* Blood products within 120 days prior to HIV screening.
* Immunoglobulin within 60 days prior to HIV screening.
* Live attenuated vaccines within 30 days prior to initial study vaccine administration.
* Investigational research agents within 30 days prior to initial study vaccine administration.
* Medically indicated subunit or killed vaccines ( e.g., influenza, pneumococcal, or allergy treatment with antigen injections) within 14 days of study vaccine administration.
* Current anti-TB prophylaxis or therapy.

Volunteer has a history of any of the following clinically significant conditions:

* Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty angioedema, or abdominal pain.
* Autoimmune disease or immunodeficiency.
* Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
* Diabetes mellitus (type I or II), with the exception of gestational diabetes.
* Thyroid disease including history of thyroidectomy and diagnoses that required medication within the past 12 months.
* Serious angioedema episodes within the previous 3 years or requiring medication in the previous 2 years.
* Hypertension that is not well controlled by medication or is more than 150/100 at enrollment.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
* Syphilis infection that is active or a positive serology due to a syphilis infection treated less than six months ago.
* Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
* Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring prolonged treatment more than 3 years ago.
* Asplenia or any condition resulting in the absence or removal of the spleen.
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment.
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgement of the investigator, would interfere with or serve as a contraindication to protocol adherence or a volunteer's ability to give informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Start 2002-10-17; Study Completion 2009-05-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Graham BS. Clinical trials of HIV vaccines. Annu Rev Med. 2002;53:207-21. doi: 10.1146/annurev.med.53.082901.104035. PMID 11818471
- [Background] Bagarazzi ML, Boyer JD, Ayyavoo V, Weiner DB. Nucleic acid-based vaccines as an approach to immunization against human immunodeficiency virus type-1. Curr Top Microbiol Immunol. 1998;226:107-43. doi: 10.1007/978-3-642-80475-5_8. No abstract available. PMID 9479839
- [Background] Heilman CA, Baltimore D. HIV vaccines--where are we going? Nat Med. 1998 May;4(5 Suppl):532-4. doi: 10.1038/nm0598supp-532. No abstract available. PMID 9585205
- [Derived] Graham BS, Koup RA, Roederer M, Bailer RT, Enama ME, Moodie Z, Martin JE, McCluskey MM, Chakrabarti BK, Lamoreaux L, Andrews CA, Gomez PL, Mascola JR, Nabel GJ; Vaccine Research Center 004 Study Team. Phase 1 safety and immunogenicity evaluation of a multiclade HIV-1 DNA candidate vaccine. J Infect Dis. 2006 Dec 15;194(12):1650-60. doi: 10.1086/509259. Epub 2006 Nov 8. PMID 17109336